CLINICAL TRIAL: NCT06391268
Title: "Investigation of the Effect of Self-Applied Emotional Liberation Technique on Pain and Stress Levels in Fibromyalgia Patients"
Brief Title: Emotional Freedom Technique (EFT) on Pain and Stress Levels in Fibromyalgia (FMS)
Acronym: EFT-FMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Buca Seyfi Demirsoy State Hospital (Other)
Responsible Party: Principal Investigator, Fatma Çetinkaya, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FCetinkaya
Record Dates: First submitted 2023-10-08; First posted 2024-04-30 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia,; Emotional free technique; pain; stress; comfort
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Intervention Model Description: 1. Determination of Subjective Units of Discomfort (SUD) (The researcher scores the distress felt on a scale between zero and ten points).
  2. Setup (The general structure of the setup sentence is "Despite this .........., I deeply and completely accept myself.")
  3. Clicking the meridian points in sequence
  4. Nine Gamut procedure (some eye movements, mumbling and counting while clicking on the Gamut point in the hand).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The group to whichEmotional freedom technique (EFT) EFT was applied by the researcher (Experimental): Emotional Freedom Technique (EFT) works on cognitive and energetic levels. While ensuring that the individual is conscious and aware of a disturbing symptom or discomfort, selected acupuncture points are touched at the same time, creating a cognitive transition and energetic release.
  1-The group to which EFT was applied by the researcher
  Interventions: Behavioral: Emotional Freedom Technique (EFT) works on cognitive and energetic levels.
- Emotional freedom technique (EFT) for fibromyalgia -2-The group that applies EFT to itself (Experimental): Emotional Freedom Technique (EFT) works on cognitive and energetic levels. While ensuring that the individual is conscious and aware of a disturbing symptom or discomfort, selected acupuncture points are touched at the same time, creating a cognitive transition and energetic release.
  2-The group that applies EFT to itself
  Interventions: Behavioral: Emotional Freedom Technique (EFT) works on cognitive and energetic levels.
- Emotional freedom technique (EFT) for fibromyalgia -3-Control group without EFT: (No Intervention): 3-Control group without EFT: Pain, problem-stress, comfort and fibromyalgia scales were applied in 3 interviews.

INTERVENTIONS:
Behavioral: Emotional Freedom Technique (EFT) works on cognitive and energetic levels. — Emotional Freedom Technique (EFT) works on cognitive and energetic levels.
  Other Names: Emotional freedom technique (EFT) for fibromyalgia
  Arms: Emotional freedom technique (EFT) for fibromyalgia -2-The group that applies EFT to itself; The group to whichEmotional freedom technique (EFT) EFT was applied by the researcher

SUMMARY:
The main aim of the study was to investigate self-administered emotional to determine the effect of the freedom technique on pain and stress levels.

The sub-objectives of the study are as follows:

1. To determine the effect of self-administration of EFT on pain level.
2. To determine the effect of self-administered EFT on stress level.
3. To determine the effect of EFT self-administration on comfort level.

DETAILED DESCRIPTION:
HYPOTHESES OF THE RESEARCH

H 1 : Between the pain levels of patients with and without self-administered EFT there is a difference.

H 2 : There is a difference between the stress levels of patients who apply EFT to themselves and those who do not. there is a difference.

H 3 : Comfort levels of patients with and without self-administered EFT there is a difference.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of fibromyalgia
* Can speak and understand Turkish
* Have time and place orientation
* No psychiatric illness,
* No vision and hearing problems.

Exclusion Criteria:

* Unstable medical condition
* Non-cooperative individuals

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2024-10-13 (Actual)

PRIMARY OUTCOMES:
Comparison of the self-EFT group | up to 24 weeks
  Comparison of the group to which EFT was performed by the researcher, Brief Scan for Stress and Problem List to assess stress and problems (Calculated out of 10 points, cut-off point is 4), Brief Pain Invertory to assess pain: The numeric pain scale is evaluated on a scale of 0-10, with "0" representing no pain and "10" representing excruciating pain. Each item is rated on a numerical scale from 0 to 10; "0" means not affected at all, "100" means completely affected).
  At the end of the study, pain and stress scores of the two experimental groups (EFT performed by the researcher and self-administered EFT) before and after EFT were analyzed and compared.
INVESTIGATION OF THE EFFECT OF SELF-APPLIED EMOTIONAL FREEDOM TECHNIQUE ON PAIN AND STRESS LEVELS IN FIBROMYALGIA PATIENTS | INVESTIGATION OF THE EFFECT OF SELF-APPLIED EMOTIONAL FREEDOM TECHNIQUE ON PAIN AND STRESS LEVELS IN FIBROMYALGIA PATIENTS
  It was determined that there was a statistically significant difference in stress thermometer measurements in the researcher-administered EFT, Self-EFT and Control groups according to time (p<0.05). As a result, the hypotheses "H1: EFT application has an effect on the pain level of patients", "H2: EFT application has an effect on the stress level of patients", "H3: EFT application has an effect on the comfort level of patients", "H4: EFT application has an effect on the fibromyalgia level of patients" were accepted. As a result of the research, significant differences were determined in pain, stress and comfort levels in all application groups.

SECONDARY OUTCOMES:
Control grouup | up to 24 weeks
  Comparison of the control group with other experimental groups, Comparison of the group to which EFT was performed by the researcher, Brief Scan for Stress and Problem List to assess stress and problems (Calculated out of 10 points, cut-off point is 4), Brief Pain Invertory to assess pain: The numeric pain scale is evaluated on a scale of 0-10, with "0" representing no pain and "10" representing excruciating pain. Each item is rated on a numerical scale from 0 to 10; "0" means not affected at all, "100" means completely affected).
  Pain, comfort, fibromyalgia effect scale scores were calculated in the control group and compared with the experimental groups.
Control grouup | The application areas of the thesis are from non-pharmacological treatments to complementary therapies.
  Comparison of the control group with other experimental groups, Comparison of the group to which EFT was performed by the researcher, Brief Scan for Stress and Problem List to assess stress and problems (Calculated out of 10 points, cut-off point is 4), Brief Pain Invertory to assess pain: The numeric pain scale is evaluated on a scale of 0-10, with "0" representing no pain and "10" representing excruciating pain. Each item is rated on a numerical scale from 0 to 10; "0" means not affected at all, "100" means completely affected).
  Pain, comfort, fibromyalgia effect scale scores were calculated in the control group and compared with the experimental groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Buca Seyfi Demirsoy Training and Research Hospital, Izmir, Turkey (Türkiye)